CLINICAL TRIAL: NCT01379222
Title: Post Approval Study Evaluating the Long Term Safety and Effectiveness of the Endurant Stent Graft System (ENGAGE PAS)
Brief Title: Endurant Stent Graft System Post Approval Study (ENGAGE PAS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10012289
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Results first posted 2019-02-04 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: AAA; Abdominal Aortic Aneurysm; EVAR; Endovascular aneurysm repair
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ENGAGE PAS De Novo Subjects (Experimental): The Endurant Stent Graft System Bifurcated device is administered to patients diagnosed with an abdominal aortic or aortoiliac aneurysm who are considered candidates for endovascular repair, per the FDA approved Instructions For Use (IFU).
  Interventions: Device: Endurant Stent Graft System

INTERVENTIONS:
Device: Endurant Stent Graft System — The Endurant Stent Graft System is designed to treat infrarenal abdominal aortic aneurysms using an endovascular approach. When placed within the aneurysm, the Endurant Stent Graft is designed to provide a permanent, alternative conduit for blood flow within the patient's vasculature by excluding the aneurysmal sac from blood flow and pressure.

SUMMARY:
The purpose of the study is to demonstrate the long term safety and effectiveness of the Endurant Stent Graft System for the endovascular treatment of infrarenal abdominal aortic aneurysms in a post-approval environment, through the endpoints established in this protocol.

The clinical objective of the study is to evaluate the long term safety and effectiveness of the Endurant Stent Graft System assessed at 5 years through freedom from Aneurysm-Related Mortality (ARM).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Indication for elective surgical repair of abdominal aortic aneurysm (AAA) with an endovascular stent graft in accordance with the applicable guidelines on endovascular interventions and the Instructions for Use of the Endurant Stent Graft System
* Signed consent form. The subject or legal representative has been informed of the nature of the trial and has consented to participate and authorized the collection and release of his medical information
* Intention to electively implant the Endurant Stent Graft System
* Ability and willingness to comply with the Clinical Investigational Plan (CIP).

Exclusion Criteria:

* High probability of non-adherence to physician's follow-up requirements
* Current participation in a concurrent trial which may confound study results
* Female of childbearing potential in whom pregnancy cannot be excluded or who is lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2011-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Schermerhorn, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (24):
- United States (24):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Stanford Hospital & Clinics, Stanford, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Bayfront Medical Center, St. Petersburg, Florida
  - Medical Center of Central Georgia (MCCG), Macon, Georgia
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Morristown Memorial Hospital, Morristown, New Jersey
  - WakeMed Health & Hospitals, Raleigh, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - The Christ Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - University of Pittsburgh Medical Center UPMC Shadyside, Pittsburgh, Pennsylvania
  - Physicians Regional Medical Center, Knoxville, Tennessee
  - Parkwest Medical Center, Knoxville, Tennessee
  - Baylor Jack and Jane Hamilton Heart and Vascular Hospital, Dallas, Texas
  - CHI Saint Luke's Health - Baylor Saint Luke's Medical Center, Houston, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ENGAGE PAS De Novo Subjects: The Endurant Stent Graft System Bifurcated device is administered to patients diagnosed with an abdominal aortic or aortoiliac aneurysm who are considered candidates for endovascular repair, per the FDA approved Instructions For Use (IFU).
  >
  > Endurant Stent Graft System: The Endurant Stent Graft System is designed to treat infrarenal abdominal aortic aneurysms using an endovascular approach. When placed within the aneurysm, the Endurant Stent Graft is designed to provide a permanent, alternative conduit for blood flow within the patient's vasculature by excluding the aneurysmal sac from blood flow and pressure.
Period: Overall Study
Arm/Group | ENGAGE PAS De Novo Subjects
Started | 178
Completed | 105
Not Completed | 73

BASELINE CHARACTERISTICS:
Arm/Group | ENGAGE PAS De Novo Subjects
Number analyzed (Participants) | 178
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 146
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 169
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 178

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Aneurysm-related Mortality Rate (ARM) at 5 Years (1826 Days)
Description: Aneurysm-Related Mortality (ARM) is defined as death from rupture of the abdominal aortic aneurysm or from any procedure intended to treat the Abdominal Aortic Aneurysm (AAA). If a death occurred within 30 days of any procedure intended to treat the AAA, then it is presumed to be aneurysm related unless there is evidence to the contrary. Deaths occurring after 30 days of any procedure intended to treat the AAA that are procedure-related should be aneurysm related.
  > All deaths will be adjudicated by a Clinical Events Committee (CEC) to determine device, procedure and/or AAA relatedness.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: Proportion of Surviving
Arm/Group | ENGAGE PAS De Novo Subjects
Number analyzed (Participants) | 178
Proportion of Surviving | 0.989 [0.973 to 1.000]

ADVERSE EVENTS:
Time Frame: 5 Years
Groups:
- 1. Engage PAS: Medtronic Engage PAS De Novo Subjects
Arm/Group | 1. Engage PAS
All-Cause Mortality (participants affected / at risk) | 48/178
Serious Adverse Events (participants affected / at risk) | 86/178
Other Adverse Events (participants affected / at risk) | 15/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Engage PAS (N=178)
Anaemia (Blood and lymphatic system disorders) | 4 (5)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Red Blood Cell Abnormality (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Arrhythmia (Cardiac disorders) | 5 (5)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Cardiac Arrest (Cardiac disorders) | 7 (7)
Cardiac Failure Congestive (Cardiac disorders) | 5 (6)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 3 (3)
Cardiopulmonary Failure (Cardiac disorders) | 3 (4)
Cardiovascular Disorder (Cardiac disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 15 (16)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Necrosis (Gastrointestinal disorders) | 1 (1)
Intestinal Ischaemia (Gastrointestinal disorders) | 2 (2)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Death (General disorders) | 3 (3)
Generalised Oedema (General disorders) | 1 (1)
Multi-Organ Failure (General disorders) | 2 (2)
Pyrexia (General disorders) | 5 (5)
Stent-Graft Endoleak (General disorders) | 6 (6)
Thrombosis In Device (General disorders) | 2 (2)
Unevaluable Event (General disorders) | 3 (3)
Cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 4 (5)
Urinary Tract Infection (Infections and infestations) | 4 (5)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 (2)
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 3 (4)
Blood Creatinine Increased (Investigations) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Balance Disorder (Nervous system disorders) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 7 (7)
Dementia (Nervous system disorders) | 1 (1)
Hepatic Encephalopathy (Nervous system disorders) | 1 (1)
Metabolic Encephalopathy (Nervous system disorders) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 2 (2)
Renal Artery Occlusion (Renal and urinary disorders) | 1 (1)
Renal Artery Stenosis (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 10 (11)
Renal Failure Acute (Renal and urinary disorders) | 1 (1)
Renal Infarct (Renal and urinary disorders) | 2 (2)
Renal Tubular Necrosis (Renal and urinary disorders) | 1 (1)
Scrotal Oedema (Reproductive system and breast disorders) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 16 (18)
Tracheal Mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic Dissection (Vascular disorders) | 1 (1)
Arterial Haemorrhage (Vascular disorders) | 1 (1)
Arterial Occlusive Disease (Vascular disorders) | 2 (2)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 4 (4)
Intermittent Claudication (Vascular disorders) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 1 (1)
Shock Haemorrhagic (Vascular disorders) | 2 (2)
Thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. Engage PAS (N=178)
Pyrexia (General disorders) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2013-06-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT01379222/Prot_000.pdf
  • Statistical Analysis Plan (2011-07-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT01379222/SAP_001.pdf